CLINICAL TRIAL: NCT07331987
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Clinical Efficacy and Safety of Probiotics in Participants With Anxiety Depression
Brief Title: Efficacy and Safety of Probiotics for Anxiety Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Moon (Guangzhou) Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MN-MOOD-102
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Anxiety Depression
Keywords: Depression; Anxiety; Mood; Probiotics
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Probiotics; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo + Escitalopram (Placebo Comparator)
  Interventions: Drug: Placebo; Combination Product: Escitalopram
- Probiotics + Escitalopram (Experimental)
  Interventions: Drug: Probiotic; Combination Product: Escitalopram

INTERVENTIONS:
Drug: Probiotic — Participants receive Probiotic product once daily by oral, 60B CFU/day for 3 months.
  Arms: Probiotics + Escitalopram
Drug: Placebo — Participants receive Placebo once daily by oral for 3 months.
  Arms: Placebo + Escitalopram
Combination Product: Escitalopram — Participants receive Escitalopram Oxalate Tablets once daily by oral, 10mg/day for 3 months.

SUMMARY:
This randomized, double-blind, placebo-controlled study will enroll 60 individuals with mild-to-moderate anxiety depression. Following a 3-month intervention and a 1-month follow-up period, the study aims to: 1) evaluate the efficacy of probiotics by comparing anxiety, depression, and sleep scores to baseline; and 2) investigate the safety and underlying mechanisms by analyzing changes in serum biomarkers, gut microbiota, and related metabolites.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age: 18-60 years old; Gender: male or female.
* 2) Meets the diagnostic criteria of Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) for a mild-to-moderate depressive or anxiety symptoms.
* 3) Hamilton Depression Rating Scale (HAM-D-24) score ≥ 8 or Hamilton Anxiety Rating Scale (HAM-A-14) score ≥ 7 at screening.
* 4) Has no used of anxiolytic or antidepressant medications (including traditional Chinese patent medicines), with the exception of Escitalopram Oxalate, within 2 weeks prior to the first dose.
* 5) For participants of childbearing potential (male or female): Must agree to use least one medically approve form of contraception (e.g., intrautering device [IUD], oral contraceptives, or condoms) throughout the trial. For female participants of childbearing potential: Must have a negative urine pregnancy test at screening and must be non-lactating.
* 6) The participant is willing and be able to provide written informed consent to participate in the study.

Exclusion Criteria:

* 1) HAM-D-24 score ≥ 35 or HAM-A-14 score ≥ 29.
* 2) Presence of significant suicidal ideation.
* 3) History or current diagnosis of neuropsychiatric disorders such as schizophrenia or epilepsy.
* 4) History of head trauma (with loss of consciousness for >10 minutes), other unstable major somatic diseases, or any somatic condition that could cause psychiatric symptoms.
* 5) Suspected intellectual disability.
* 6) History of alcohol or substance abuse prior to enrollment.
* 7) Cranial magnetic resonance imaging (MRI) reveals organic lesions.
* 8) Participants who are deemed unsuitable for the study by the investigator for any other reason.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HAM-D-24) | Baseline, Day 30, Day 90, Day 120 (follow up)
  Depression symptoms will be assessed using the 24-item Hamilton Depression Rating Scale (HAM-D-24) at baseline and the specified time points during the study. With higher scores indicating more severe depression, and scores categorized as <8 non-depressed, 8-19 mild, 20-34 moderate, ≥35 severe for diagnosis and monitoring treatment response.
Hamilton Anxiety Rating Scale (HAM-A) | Baseline, Day 30, Day 90, Day 120 (follow up)
  Anxiety symptoms will be evaluated using 14-item Hamilton Anxiety Rating Scales (HAM-A) at baseline and the specified time point during the study. Each item is scored on a scale of 0 (not present) to 4 (severe). The total score, calculated by summing all items, ranges from 0 to 56, with higher scores indicating greater anxiety severity, where 0-7 indicates no/minimal, 8-14 mild, 15-23 moderate and ≥24 severe.

SECONDARY OUTCOMES:
The Pittsburgh Sleep Quality Index (PSQI) | Baseline, Day 30, Day 90, Day 120 (follow up)
  Assesses sleep quality from baseline to end of the study by questionnaire of The Pittsburgh Sleep Quality Index (PSQI). There are 19 items that are used to generate 7 component scores, which then are added together to determine a global score that ranges between 0 to 21, where higher scores reflect worse sleep quality.
Gastrointestinal Symptom Rating Scale (GSRS) | Baseline, Day 30, Day 90, Day 120 (follow up)
  Assessment of gastrointestinal symptoms will conducted at baseline and throughout the study period. The GSRS is a disease-specific instrument of 15 items combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided